CLINICAL TRIAL: NCT04607928
Title: Phase-II Randomized Clinical Trial to Evaluate the Effect of Pirfenidone Compared to Placebo in Post-COVID19 Pulmonary Fibrosis
Brief Title: Pirfenidone Compared to Placebo in Post-COVID19 Pulmonary Fibrosis COVID-19
Acronym: FIBRO-COVID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Maria Molina, Coordinating Investigator, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-002518-42
Record Dates: First submitted 2020-10-28; First posted 2020-10-29 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Fibrotic Pulmonary Sequelae Post-COVID19 Infection
MeSH Terms: interventions — pirfenidone

STUDY DESIGN:
Intervention Model Description: 2:1 (treatment:placebo)
Who Masked: Participant, Care Provider, Investigator
Masking Description: doble blinded, IVRSystem
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): No anti-fibrotic treatment. Patients in placebo and treatment arm may be on corticosteroid treatment
  Interventions: Drug: Placebo
- Treatment (Experimental): Pirfenidone
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Comparing the effect of pirfenidone in avoiding establishing or progression of fibrosis induced after COVID19 infection
  Arms: Treatment
Drug: Placebo — Comparing the effect of pirfenidone in avoiding establishing or progression of fibrosis induced after COVID19 infection
  Arms: Placebo

SUMMARY:
Study population: Patients with fibrotic lung sequelae after recovery from acute phase of severe COVID19 pneumonia Objectives: To evaluate the effect of pirfenidone administered for 24 weeks in patients who have pulmonary fibrotic changes after suffering severe COVID19 pneumonia, analysed by

* % change in forced vital capacity (FVC)
* % fibrosis in high resolution computed tomography (HRCT) of the lung

DETAILED DESCRIPTION:
Has been designed a clinical trial with an experimental and a control arm, with 2 experimental subjects per control (2:1), we will have to study 98 experimental subjects and 50 control subjects, in total 148 patients. Randomization will be performed using a centralized electronic system (IVRS) with 2: 1 randomized concealed assignment. This randomization will be done by permuted blocks.

The study population will be patients with fibrosing lung sequelae after recovery from severe COVID19 pneumonia.

This is a double-blind, masked, placebo-controlled clinical trial: the patient and the investigator are unaware of the assigned treatment the patient receives.

Patients will follow a total of 5 clinic visits; V0 (screening, -1 days - +42 days from signing the Informed Consent), V1 (randomization), V2 (week 12), V3 (week 24 or end of treatment), V4 (week 28 or follow-up).

Visits Plan

* V0 - Screening: Initially, the informed consent will be collected. Subsequently, we will proceed to collect clinical variables, blood tests and radiological characteristics (chest CT scan; radiological signs of fibrosis such as tractional bronchiolectasis, honeycombing, loss of lung volume and reticulation).
* V1 - Randomization: Before starting the drug:

Control analytics Serum pregnancy test for all women of childbearing age KBILD quality of life test. This validated questionnaire will be completed by the patient following the instructions of the staff.

Spirometry (CVF) and plethysmography (DLCO) TM6m. Extraction of blood for DNA isolation (in those cases that have specifically signed the IC for genetics) and proteins (serum).

Once the screening evaluation has been completed, eligibility will depend on meeting the inclusion criteria and not presenting any exclusion criteria. Those cases that are not eligible will be informed and an adequate explanation will be provided.

* V2 - 12 weeks after starting medication. The patient's clinical status will be collected
* V3 - 24 weeks (end of treatment period). Clinical data and quality of life test (KBILD) will be collected, and chest CT scan, spirometry-plethysmography and TM6m will be performed. Blood will be drawn for protein isolation (serum).
* V4 - 28 weeks (follow-up). Clinical and analytical variables will be collected.

Patients will have the telephone number of the main researcher or someone from the team where they can call 24 hours, which will be specified on the patient's card (where it will be identified that the patient participates in this study). In case of presenting any problem or side effect in the period between visits, the patient will go to the center and an additional visit will be made.

Study treatment:

Pirfenidone Name: Esbriet 267 mg hard capsules Dosage: 267 mg (capsules) Manufacturer: Roche Pharma AG

Study drug administration schedule: The study medication will be started at incremental doses, starting with 1602 mg / day (divided into three doses every 8 hours, 267 mg capsules with each meal) and, if there is no liver or associated serious events, will be increased on the 7th day to full doses of 2403 mg / day. The dose increase can be extended for one more week if the investigator considers it safer (slight elevation of liver enzymes, digestive discomfort or clear anorexia). Subsequently, 2403 mg / day will be maintained (3 capsules in each meal during the day) except if it is necessary to reduce the dose or suspend the drug due to adverse effects or associated problems (at the discretion of the researcher).

Concomitant treatments prohibited:

The use of the following therapies is prohibited during study treatment:

* Cytotoxic, immunosuppressant, cytokine modulators, including but not limited to azathioprine, bosentan, ambrisentan, cyclophosphamide, cyclosporine, etanercept, iloprost, infliximab, leukotriene antagonists, methotrexate, high doses of corticosteroids (more than 15 mg / day of prednisone or equivalent for more than 20 days), mycophenolate mofetil, tacrolimus, montelukast, tetrathiomolybdate, TNF-α inhibitors, imatinib mesylate, interferon gamma-1b, and tyrosine kinase inhibitors.
* Strong CYP1A2 inhibitors (eg, Fluvoxamine, Enoxacin), P-glycoprotein inhibitors (eg, Ketoconazole, erythromycin) or CYP3A4 (eg, Ketoconazole, erythromycin), or their inducers (eg. Eg, rifampicin, carbamazepine, phenytoin).
* Any investigational therapy in an active clinical trial.
* Because moderate CYP1A2 inhibitors (eg, Ciprofloxacin) increase the systemic exposure of pirfenidone (Esbriet® US label 2014), if ciprofloxacin is administered, it should be limited to 250 or 500 mg daily (QD), and the patient should be closely monitored.

Prohibited foods: The consumption of grapefruit juice will be prohibited during the study.

Additional restriction: The use of any form of tobacco consumption will be prohibited.

Criteria for patient withdrawal from the study Participation in the study is voluntary and the subjects can withdraw at any time without having to give explanations and without this implying a detriment to the healthcare they receive in the future.

For her part, the researcher must withdraw a subject from the study:

* Adverse event or clinical situation of the patient that, in the clinical opinion, makes it necessary to withdraw from the study. Patients can interrupt the medication for up to 14 days, returning to the previous dose without requiring titration. If they interrupt for more than 14 days, they have to gradually increase the dose. If the patient cannot tolerate the minimum dose, then the treatment will be withdrawn, allowing study visits to be completed.
* Request for withdrawal by the patient.
* Serious violation of protocol.
* Loss of follow-up.
* Pregnancy during the study. When a subject withdraws from the study, the investigator will record the reason or reasons for withdrawal in the original documents in the Medical Record.

End of clinical trial is defined as the date the last recruited patient completes the last visit (LPLV). The last patient is expected to complete the last visit 4 weeks after the last patient has completed treatment, which is expected to happen 14 months after the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Signed Informed Consent Form
* Ability to comply with the study protocol in the opinion of the Investigator
* Confirmation of SARS-COV2 infection in previous weeks (Confirmation of negativity or no activity of SARS-COV2 before randomization using the usual tests performed in the hospital), which induced severe pneumonia and ARDS, with subsequent torpid recovery and/or incipient clinical-radiological signs of pulmonary fibrosis.
* HRCT with fibrotic radiological changes of at least 5% after recovery from the acute process (HRCT chest during the screening period, performed minimum after 1 month of the acute phase and maximum 90 days after hospital discharge)
* Be able to understand the information given and sign the informed consent
* For women or men of childbearing age who are not sterile, a commitment to use non-hormonal contraception during the 24-week treatment period will be required.

Exclusion Criteria:

* Use of systemic steroids (oral or intravenous) at doses greater than 15 mg/day one month prior to randomisation.
* Severe or moderate myopathy that may associate a decrease of FVC.
* Severe or life-limiting chronic disease prior to COVID19 infection, including severe asthma, cancer, clinical dementia, IPF, or uncontrolled ischemic cardiomyopathy.
* Treatment with pirfenidone or nintedanib prior to Covid19
* Concomitant treatment with significant interactions with pirfenidone (such as fluvoxamine).
* Participation in any other investigational trial throughout the study
* Active smoking.
* Relevant blood alterations in the analysis made during the screening period:

  * Total bilirubin > 2 ULN
  * AST/SGOT or ALT/SGPT > 2.5 ULN
  * Alkaline phosphatase >3.0 ULN
  * Creatinine Clearance <40 mL/min, calculated by the Cockcroft-Gault formula
* Pregnancy or lactation
* Concomitant treatments that can cause severe digestive problems.
* Gastric surgery in the last 3 months or similar procedures that may increase gastric intolerance.
* Inability to complete required visits.
* Previous intolerance or allergy to pirfenidone or hypersensitivity to any of its excipients.
* History of angioedema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
To investigate the effect of pirfenidone on fibrotic signs induced by COVID19 infection | 24 weeks
  To investigate the effect of pirfenidone administered for 24 weeks measuring the number of patients who have pulmonary fibrotic changes from baseline after suffering severe COVID19 pneumonia, analysed by
  * Change From Baseline in % in forced vital capacity (FVC)
  * Change From Baseline % fibrosis in high resolution computed tomography (HRCT) of the lung

SECONDARY OUTCOMES:
Maintenance of stability or functional improvement FVC | 24 weeks
  Number of patients who show maintenance of stability or functional improvement: stability will be considered when the FVC does not increase more than 10% or does not decrease more than 10% and the DLCO does not increase more than 15% or decreases more than 15%. An increase in% FVC greater than 10% or in DLCO greater than 15% will be considered significant improvement.
Decreased oxygen requirement for physical activity | 24 weeks
  Rate of decreased oxygen requirement for physical activity in patients
Improved exercise capacity (> 50 meter improvement or less decrease in% oxygen saturation) in the TM6m | 24 weeks
  Number of patients who have improved exercise capacity (> 50 meter improvement or less decrease in% oxygen saturation) in the TM6m
Hospitalizations (general and due to respiratory problems) | 24 weeks
  Number of Hospitalizations (general and due to respiratory problems)
Visits to the Emergency or Day Hospital for respiratory causes | 24 weeks
  Number of Visits to the Emergency or Day Hospital for respiratory causes
Lung transplantation | 24 weeks
  Number of patients who need Lung transplantation
Death | 24 weeks
  Number of patients who die

CONTACTS AND LOCATIONS:
Overall Officials: Maria Molina-Molina, MD, PhD, Study Chair — Institut d'Investigació Biomèdica de Bellvitge
Locations (8):
- Spain (8):
  - University Hospital of Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clínic, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital La Princes, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No